CLINICAL TRIAL: NCT03905798
Title: LORA-PITA (REGISTERED) Intravenous Injection 2 mg General Investigation
Brief Title: LORA-PITA IV General Investigation
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3541003; NCT03905798 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Status Epilepticus
Keywords: Status Epilepticus;; Lorazepam;; LORA-PITA;; Ativan
MeSH Terms: conditions — Status Epilepticus | interventions — Lorazepam

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lorazepam: Patients administered Lorazepam in accordance with the indication (for Status Epilepticus, SE) and have no history of using this drug
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Lorazepam — The usual dose of lorazepam in adults is 4 mg administered intravenously. The drug should be given slowly with the administration rate at 2 mg/min as a guide. If necessary, 4 mg may be added but the dose should not exceed 8 mg as the sum of initial and additional doses.
  The usual dose of lorazepam in children aged 3 months or older is 0.05 mg/kg (up to 4 mg) administered intravenously. The drug should be given slowly with the administration rate at 2 mg/min as a guide. If necessary, 0.05 mg/kg may be added but the dose should not exceed 0.1 mg/kg as the sum of initial and additional doses.
  Other Names: LORA-PITA

SUMMARY:
Secondary Data Collection:To confirm the effectiveness and safety profiles under the actual medical practice of LORA-PITA in Japan.

DETAILED DESCRIPTION:
To confirm the effectiveness and safety profiles under the actual medical practice of LORA-PITA for Status Epilepticus patients in Japan.

ELIGIBILITY:
Inclusion Criteria: Patients administered Lorazepam in accordance with the indication (for Status Epilepticus) and have no history of using this drug.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients administered Lorazepam in accordance with the indication (for Status Epilepticus) and have no history of using this drug.
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Local Country office, Tokyo, Shibuya-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3541003

RESULTS

PARTICIPANT FLOW:
Groups:
- LORA-PITA Intravenous Injection 2mg (Lorazepam): This study was conducted by fixed-point all participants surveillance system in participants who received LORA-PITA as indicated in the approved local product document. The observation period was from the first dose received to 24 hours after the last dose received. A follow-up period was 24 hours after the end of the last dose, and if the follow-up period was less than 24 hours, such participants were deemed as withdrawals.
  The pediatric (< 16 years) and adult (≥ 16 years) participants' initial doses were 0.25 to 4.00 mg (0.025 to 0.098 mg/kg) and 1.50 to 4.00 mg, respectively. The pediatric and adult participants' second doses were 0.40 to 2.00 mg (0.024 to 0.050 mg/kg) and 2.00 to 4.00 mg, respectively. The pediatric and adult participants' third doses were 0.80 mg (0.024 mg/kg) and 2.00 to 4.00 mg, respectively.
Period: Overall Study
Arm/Group | LORA-PITA Intravenous Injection 2mg (Lorazepam)
Started | 206
Completed | 112
Not Completed | 94
Not completed — No informed consent for notification/publication of study results | 94

BASELINE CHARACTERISTICS:
Population: A total of 112 participants completed the study. There were no cases excluded from the safety analysis set, and all 112 cases were included in the safety analysis population.
Arm/Group | LORA-PITA Intravenous Injection 2mg (Lorazepam)
Number analyzed (Participants) | 112
Age, Customized [Number; unit: Participants]
  <16 years | 23
  ≥16 and <65 years | 40
  ≥65 years | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of the Participants With Adverse Drug Reactions
Description: An adverse drug reaction (ADR) was a treatment-related adverse event, and any untoward medical occurrence attributed to LORA-PITA in a participant who received LORA-PITA. A serious adverse drug reaction (SADR) was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Relatedness to LORA-PITA was assessed by the physician.
Time Frame: From the first dose of LORAPITA to 24 hours after the end of the last dose, up to approximately 2 days.
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received LORA-PITA at least once. Participants without informed consent for notification/publication of study results were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | LORA-PITA Intravenous Injection 2mg (Lorazepam)
Number analyzed (Participants) | 112
Participants | 7

2. Secondary Outcome: Proportion of Participants Whose Initial Seizure Stopped Within 10 Minutes After the Administration of Final Dose and Who Continued Seizure-free for at Least 30 Minutes (Participants in Whom LORA-PITA Was Used as the First-line Treatment)
Description: Epileptic seizures subject to treatment with LORA-PITA were evaluated as effectiveness evaluation.
  Definition of responders to the first or second administration of LORA-PITA: A responder was defined as a participant whose seizure resolved within 10 minutes after the first administration of LORA-PITA or the second administration (10 to 30 minutes after the first administration) and who did not require additional treatment with other drugs for the target disease within 30 minutes after the end of administration (excluding prophylactic administration) and had no recurrent seizure.
Time Frame: From the first dose of LORAPITA to 24 hours after the end of the last dose, up to approximately 2 days.
Population: The efficacy analysis set (84 participants) comprised of participants in the safety analysis set in whom LORA-PITA was used as the first-line treatment with evaluable effectiveness, excluding participants who met any of the following conditions: effectiveness evaluation has not been reported at all or the administration was as the second-line treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LORA-PITA Intravenous Injection 2mg (Lorazepam)
Number analyzed (Participants) | 84
Percentage of Participants | 64.3 [53.1 to 74.4]

3. Secondary Outcome: Proportion of Participants Whose Initial Seizure Stopped Within 10 Minutes After the Administration of Final Dose and Who Continued Seizure-free for at Least 30 Minutes (Efficacy Analysis Set)
Description: as for outcome 2
Time Frame: From the first dose of LORAPITA to 24 hours after the end of the last dose, up to approximately 2 days.
Population: The efficacy analysis set (104 participants) comprised of participants in the safety analysis set in whom LORA-PITA was used and had evaluable effectiveness data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LORA-PITA Intravenous Injection 2mg (Lorazepam)
Number analyzed (Participants) | 104
Percentage of Participants | 62.5 [52.5 to 71.8]

ADVERSE EVENTS:
Time Frame: From the first dose of LORAPITA to 24 hours after the end of the last dose, up to approximately 2 days.
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | LORA-PITA Intravenous Injection 2mg (Lorazepam)
All-Cause Mortality (participants affected / at risk) | 0/112
Serious Adverse Events (participants affected / at risk) | 1/112
Other Adverse Events (participants affected / at risk) | 9/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LORA-PITA Intravenous Injection 2mg (Lorazepam) (N=112)
Ventricular tachycardia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LORA-PITA Intravenous Injection 2mg (Lorazepam) (N=112)
Bradycardia (Cardiac disorders) | 1
Blood pressure decreased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Renal impairment (Renal and urinary disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT03905798/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT03905798/SAP_001.pdf